CLINICAL TRIAL: NCT02573779
Title: Intestinal Microbiota and Short Term Outcomes in Very Low Birth Weight Infants Fed Primarily Donor Human Milk Compared to Infants Fed Primarily Mother's Own Milk
Brief Title: Growth and Microbiome Development in Very Low Birth Weight Infants Fed Primarily Mother's Own Milk vs. Donor Human Milk
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Amy Hair, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-36828
Record Dates: First submitted 2015-10-08; First posted 2015-10-12 (Estimated); Results first posted 2020-04-29 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Infant, Very Low Birth Weight
Keywords: human milk; enteral nutrition; microbiome; microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At time of initial consent for the study, mothers will also be asked for consent to obtain a small sample (0.2-0.5 mL) of colostrum or expressed milk produced in the first week of life, as well as weekly milk samples thereafter, in order to analyze bacterial content of milk as it compares to the developing infant microbiome. For infants who receive primarily donor milk, weekly samples of the milk they receive may similarly be analyzed for bacterial content.
  Infant stool samples will be collected during the first week of life and then at weekly intervals for six weeks. The samples will be analyzed via 16S rRNA sequencing to determine diversity of intestinal microbiota. Additional analysis for metabolomics will be considered if lab availability and cost allows.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Infants fed mother's own milk: Infants fed >50% mother's own milk with enteral feeding.
  Interventions: Other: Observational - no intervention
- Donor milk fed infants: Infants fed <50% mother's own milk (and thus >50% donor human milk) with enteral feeding.
  Interventions: Other: Observational - no intervention

INTERVENTIONS:
Other: Observational - no intervention — This study will observe cohorts of infants who are fed primarily either their own mother's milk or donor milk as part of their routine care. No direct intervention is performed as part of the study.

SUMMARY:
A study to compare growth, development of the intestinal bacterial environment, and other short term outcomes in groups of babies fed primarily their own mother's milk compared to those who receive primarily donor human milk. The investigators hypothesize that infants who receive primarily their own mother's milk will have better growth, a more diverse intestinal bacterial environment, and possibly some improved short term outcomes such as better feeding tolerance and lower rates of infection.

DETAILED DESCRIPTION:
Background: Human milk feeding provides numerous benefits to preterm infants due to improvements in gastrointestinal maturation, host defense, infection rates, and improved long-term outcomes in neurodevelopment as well as cardiovascular and metabolic disease. There is accumulating evidence that an exclusive human milk-based diet decreases the rates of necrotizing enterocolitis (NEC) and death, and is associated with better feeding tolerance in very low birth weight (VLBW) infants than a diet of bovine milk-based products. In order to provide VLBW infants the benefits afforded by human milk feeding, the use of donor milk (DM) in neonatal intensive care units (NICU) has increased as many mothers are unable to provide sufficient milk needed for their premature infants. While there have been numerous studies that have favorably compared feeding of mother's own milk (MOM) to formula as well as studies that compare DM to formula, there are relatively few that compare maternal milk to donor milk.

In regard to feeding tolerance and infection prevention, it has been proposed that DM may be less beneficial than MOM due to reduction in biologically active components during pasteurization, including human milk oligosaccharides (HMOs) and other immunological factors, growth factors, and hormones. Finally, alterations in the intestinal microbiota of preterm infants are suspected to contribute to disease states such as NEC, specifically within infants who have decreased microbial diversity. To the investigators knowledge, no studies comparing the intestinal microbiota among infants fed primarily MOM versus those fed primarily DM have been published.

Purpose: To compare growth velocities, time to reach full enteral feeding volume, intestinal microbiota, and short term outcomes (NEC, late-onset sepsis, white matter injury) between infants fed primarily mother's own milk versus pasteurized donor human milk.

Hypothesis: Infants fed primarily (50% or greater) mother's own milk will have increased intestinal microbiome diversity compared to infants fed primarily pasteurized donor human milk.

Design: This prospective cohort study will be conducted in the Level III NICU at Texas Children's Hospital - Pavilion for Women and the Level II NICU at Texas Children's Hospital -- West Tower. Infants less than 1500 g birth weight will be fed exclusively human milk (mother's milk and or donor breast milk) fortified with donor human milk-derived fortifier per the investigators hospital guidelines. Once enteral feeding is established, infants will be categorized into cohorts based on percentage of feeding volume consisting of mother's own milk, including broad categorization of greater than 50% maternal milk versus less than 50%, and possibly tiered analysis of infants who receive less 25% maternal milk, 25-75% maternal milk, and greater than 75% maternal milk.

An enrollment goal of greater than 125 infants including twins and multiples will be targeted for adequate sample size.

Procedure: Infants will be enrolled within 72 hours of birth and started on parenteral nutrition and enteral human milk feedings per standardized feeding protocols and discretion of the attending neonatologist on service. Decisions to decrease or discontinue enteral feedings due to medical instability will be made by the attending neonatologist. Infants will be preferentially fed their own mothers' milk when available. For mothers who are unable to express adequate milk volume for their infants, pooled, pasteurized donor human milk will be offered per established NICU protocol. Feeds will be supplemented with human-milk based fortifier per protocol.

At time of initial consent for the study, mothers will also be asked for consent to obtain a small sample (0.2-0.5 mL) of colostrum or expressed milk produced in the first week of life, as well as weekly milk samples thereafter, in order to analyze bacterial content of milk as it compares to the developing infant microbiome. However, consent for milk collection is not required for the infant's participation in the study. For infants who receive primarily donor milk, weekly samples of the milk they receive may similarly be analyzed for bacterial content.

Infant stool samples will be collected during the first week of life and then at weekly intervals for six weeks for research purposes. The samples will be analyzed via 16S rRNA sequencing to determine diversity of intestinal microbiota. Additional analysis for metabolomics will be considered if lab availability and cost allows.

Once weekly, a research nurse or physician will document growth measurements, including weight, length, and head circumference. Outcome data from the infants' medical records will be recorded, including time to regain birth weight, feeding tolerance as indicated by time required to reach full enteral feeding volumes of 100 ml/kg/day (for hydration) and 130-160 ml/kg/day (final goal volume for nutrition), and rates of NEC, spontaneous intestinal perforation (SIP), late-onset sepsis, and bronchopulmonary dysplasia (BPD). As all preterm infants less than 1000 g birth weight born at TCH-PFW have routinely performed brain MRIs at term gestation or hospital discharge, enrolled infants who fall into this subgroup will have their MRI results reviewed for outcome analysis.

Additional medical record data for collection will include mechanism of delivery (cesarean vs. vaginal), antibiotics received by mother during 2nd and 3rd trimester as well as at time of delivery and while nursing/expressing milk, antibiotics received by baby during hospitalization, length of hospitalization, postmenstrual age at discharge, days NPO, days of parenteral nutrition, percentage of patients with patent ductus arteriosus, and rates of intraventricular hemorrhage, retinopathy of prematurity, and death.

Although there is no long-term follow up currently designed for this study, at time of initial enrollment there will be an optional consent to allow study personnel to access medical records for patients who go on to have neurodevelopmental follow up visits at clinics within the investigators institution. There will also be optional consent for families to be contacted when the infant is approximately 6, 12, 18, and 24 months for developmental follow up. This will allow for possible comparison of neurodevelopmental outcomes at approximately 18-24 months in the subgroup of patients whose mothers consent to these aspects of the study.

No labs will be requested for research purposes. No interventions are part of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Infants less than 72 hours old and less than 1500 g birth weight, who have reasonable expectation of survival and can adhere to a feeding protocol involving mother's own milk and/or donor milk that will include fortification using Prolacta and potentially human cream.

Exclusion Criteria:

* Exclusion criteria will include birth weight greater than 1500 g, age > 72 hours old, major congenital anomalies, clinically significant heart disease, abdominal wall defects and/or intestinal atresias, severe perinatal hypoxia, or otherwise less than reasonable expectation of survival through the study period.

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn infants less than 1500 g birth weight who are fed primarily either mother's own milk or donor human milk.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Hair, MD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital
Locations (2):
- United States (2):
  - Baylor College of Medicine / Texas Children's Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Background] Schanler RJ. Outcomes of human milk-fed premature infants. Semin Perinatol. 2011 Feb;35(1):29-33. doi: 10.1053/j.semperi.2010.10.005. PMID 21255704
- [Background] Sullivan S, Schanler RJ, Kim JH, Patel AL, Trawoger R, Kiechl-Kohlendorfer U, Chan GM, Blanco CL, Abrams S, Cotten CM, Laroia N, Ehrenkranz RA, Dudell G, Cristofalo EA, Meier P, Lee ML, Rechtman DJ, Lucas A. An exclusively human milk-based diet is associated with a lower rate of necrotizing enterocolitis than a diet of human milk and bovine milk-based products. J Pediatr. 2010 Apr;156(4):562-7.e1. doi: 10.1016/j.jpeds.2009.10.040. Epub 2009 Dec 29. PMID 20036378
- [Background] Cristofalo EA, Schanler RJ, Blanco CL, Sullivan S, Trawoeger R, Kiechl-Kohlendorfer U, Dudell G, Rechtman DJ, Lee ML, Lucas A, Abrams S. Randomized trial of exclusive human milk versus preterm formula diets in extremely premature infants. J Pediatr. 2013 Dec;163(6):1592-1595.e1. doi: 10.1016/j.jpeds.2013.07.011. Epub 2013 Aug 20. PMID 23968744
- [Background] Abrams SA, Schanler RJ, Lee ML, Rechtman DJ. Greater mortality and morbidity in extremely preterm infants fed a diet containing cow milk protein products. Breastfeed Med. 2014 Jul-Aug;9(6):281-5. doi: 10.1089/bfm.2014.0024. Epub 2014 May 27. PMID 24867268
- [Background] Sisk PM, Lovelady CA, Gruber KJ, Dillard RG, O'Shea TM. Human milk consumption and full enteral feeding among infants who weigh </= 1250 grams. Pediatrics. 2008 Jun;121(6):e1528-33. doi: 10.1542/peds.2007-2110. PMID 18519456
- [Background] Schanler RJ, Shulman RJ, Lau C. Feeding strategies for premature infants: beneficial outcomes of feeding fortified human milk versus preterm formula. Pediatrics. 1999 Jun;103(6 Pt 1):1150-7. doi: 10.1542/peds.103.6.1150. PMID 10353922
- [Background] Section on Breastfeeding. Breastfeeding and the use of human milk. Pediatrics. 2012 Mar;129(3):e827-41. doi: 10.1542/peds.2011-3552. Epub 2012 Feb 27. PMID 22371471
- [Background] Schanler RJ. Mother's own milk, donor human milk, and preterm formulas in the feeding of extremely premature infants. J Pediatr Gastroenterol Nutr. 2007 Dec;45 Suppl 3:S175-7. doi: 10.1097/01.mpg.0000302967.83244.36. PMID 18185087
- [Background] Hair AB, Hawthorne KM, Chetta KE, Abrams SA. Human milk feeding supports adequate growth in infants </= 1250 grams birth weight. BMC Res Notes. 2013 Nov 13;6:459. doi: 10.1186/1756-0500-6-459. PMID 24220185
- [Background] Hair AB, Blanco CL, Moreira AG, Hawthorne KM, Lee ML, Rechtman DJ, Abrams SA. Randomized trial of human milk cream as a supplement to standard fortification of an exclusive human milk-based diet in infants 750-1250 g birth weight. J Pediatr. 2014 Nov;165(5):915-20. doi: 10.1016/j.jpeds.2014.07.005. Epub 2014 Aug 15. PMID 25130571
- [Background] Dewey KG, Heinig MJ, Nommsen-Rivers LA. Differences in morbidity between breast-fed and formula-fed infants. J Pediatr. 1995 May;126(5 Pt 1):696-702. doi: 10.1016/s0022-3476(95)70395-0. PMID 7751991
- [Background] Le Huerou-Luron I, Blat S, Boudry G. Breast- v. formula-feeding: impacts on the digestive tract and immediate and long-term health effects. Nutr Res Rev. 2010 Jun;23(1):23-36. doi: 10.1017/S0954422410000065. Epub 2010 May 10. PMID 20450531
- [Background] Duijts L, Ramadhani MK, Moll HA. Breastfeeding protects against infectious diseases during infancy in industrialized countries. A systematic review. Matern Child Nutr. 2009 Jul;5(3):199-210. doi: 10.1111/j.1740-8709.2008.00176.x. PMID 19531047
- [Background] ESPGHAN Committee on Nutrition; Arslanoglu S, Corpeleijn W, Moro G, Braegger C, Campoy C, Colomb V, Decsi T, Domellof M, Fewtrell M, Hojsak I, Mihatsch W, Molgaard C, Shamir R, Turck D, van Goudoever J. Donor human milk for preterm infants: current evidence and research directions. J Pediatr Gastroenterol Nutr. 2013 Oct;57(4):535-42. doi: 10.1097/MPG.0b013e3182a3af0a. PMID 24084373
- [Background] Bertino E, Giuliani F, Baricco M, Di Nicola P, Peila C, Vassia C, Chiale F, Pirra A, Cresi F, Martano C, Coscia A. Benefits of donor milk in the feeding of preterm infants. Early Hum Dev. 2013 Oct;89 Suppl 2:S3-6. doi: 10.1016/j.earlhumdev.2013.07.008. Epub 2013 Aug 6. PMID 23932110
- [Background] Quigley M, McGuire W. Formula versus donor breast milk for feeding preterm or low birth weight infants. Cochrane Database Syst Rev. 2014 Apr 22;(4):CD002971. doi: 10.1002/14651858.CD002971.pub3. PMID 24752468
- [Background] Schanler RJ, Lau C, Hurst NM, Smith EO. Randomized trial of donor human milk versus preterm formula as substitutes for mothers' own milk in the feeding of extremely premature infants. Pediatrics. 2005 Aug;116(2):400-6. doi: 10.1542/peds.2004-1974. PMID 16061595
- [Background] Montjaux-Regis N, Cristini C, Arnaud C, Glorieux I, Vanpee M, Casper C. Improved growth of preterm infants receiving mother's own raw milk compared with pasteurized donor milk. Acta Paediatr. 2011 Dec;100(12):1548-54. doi: 10.1111/j.1651-2227.2011.02389.x. Epub 2011 Jul 14. PMID 21707744
- [Background] Garcia-Lara NR, Vieco DE, De la Cruz-Bertolo J, Lora-Pablos D, Velasco NU, Pallas-Alonso CR. Effect of Holder pasteurization and frozen storage on macronutrients and energy content of breast milk. J Pediatr Gastroenterol Nutr. 2013 Sep;57(3):377-82. doi: 10.1097/MPG.0b013e31829d4f82. PMID 23752081
- [Background] Marx C, Bridge R, Wolf AK, Rich W, Kim JH, Bode L. Human milk oligosaccharide composition differs between donor milk and mother's own milk in the NICU. J Hum Lact. 2014 Feb;30(1):54-61. doi: 10.1177/0890334413513923. Epub 2013 Nov 26. PMID 24282194
- [Background] Evans TJ, Ryley HC, Neale LM, Dodge JA, Lewarne VM. Effect of storage and heat on antimicrobial proteins in human milk. Arch Dis Child. 1978 Mar;53(3):239-41. doi: 10.1136/adc.53.3.239. PMID 306224
- [Background] Torrazza RM, Neu J. The altered gut microbiome and necrotizing enterocolitis. Clin Perinatol. 2013 Mar;40(1):93-108. doi: 10.1016/j.clp.2012.12.009. PMID 23415266
- [Background] Wang Y, Hoenig JD, Malin KJ, Qamar S, Petrof EO, Sun J, Antonopoulos DA, Chang EB, Claud EC. 16S rRNA gene-based analysis of fecal microbiota from preterm infants with and without necrotizing enterocolitis. ISME J. 2009 Aug;3(8):944-54. doi: 10.1038/ismej.2009.37. Epub 2009 Apr 16. PMID 19369970
- [Background] Mai V, Young CM, Ukhanova M, Wang X, Sun Y, Casella G, Theriaque D, Li N, Sharma R, Hudak M, Neu J. Fecal microbiota in premature infants prior to necrotizing enterocolitis. PLoS One. 2011;6(6):e20647. doi: 10.1371/journal.pone.0020647. Epub 2011 Jun 6. PMID 21674011
- [Background] Harmsen HJ, Wildeboer-Veloo AC, Raangs GC, Wagendorp AA, Klijn N, Bindels JG, Welling GW. Analysis of intestinal flora development in breast-fed and formula-fed infants by using molecular identification and detection methods. J Pediatr Gastroenterol Nutr. 2000 Jan;30(1):61-7. doi: 10.1097/00005176-200001000-00019. PMID 10630441
- [Background] Hanson LA, Korotkova M, Telemo E. Breast-feeding, infant formulas, and the immune system. Ann Allergy Asthma Immunol. 2003 Jun;90(6 Suppl 3):59-63. doi: 10.1016/s1081-1206(10)61662-6. PMID 12839115
- [Background] Ward RE, Ninonuevo M, Mills DA, Lebrilla CB, German JB. In vitro fermentation of breast milk oligosaccharides by Bifidobacterium infantis and Lactobacillus gasseri. Appl Environ Microbiol. 2006 Jun;72(6):4497-9. doi: 10.1128/AEM.02515-05. PMID 16751577
- [Background] Bjorkstrom MV, Hall L, Soderlund S, Hakansson EG, Hakansson S, Domellof M. Intestinal flora in very low-birth weight infants. Acta Paediatr. 2009 Nov;98(11):1762-7. doi: 10.1111/j.1651-2227.2009.01471.x. Epub 2009 Aug 8. PMID 19673724
- [Derived] Ford SL, Lohmann P, Preidis GA, Gordon PS, O'Donnell A, Hagan J, Venkatachalam A, Balderas M, Luna RA, Hair AB. Improved feeding tolerance and growth are linked to increased gut microbial community diversity in very-low-birth-weight infants fed mother's own milk compared with donor breast milk. Am J Clin Nutr. 2019 Apr 1;109(4):1088-1097. doi: 10.1093/ajcn/nqz006. PMID 30982856

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible study participants included premature inborn infants at <1500 g BW with no barriers to enteral milk feeding. Infants were approached and enrolled within the first 72 hr of life.
Pre-assignment Details: Of 223 inborn infants <1500 g BW between September 2015 to August 2016, 33 infants were excluded, 59 could not be enrolled within 72 h, and 6 were not enrolled because their parents declined. Of the 125 enrolled infants, 8 were removed from the study owing to GI defects or complications unknown at time of enrollment that precluded enteral feeding.
Period: Overall Study
Arm/Group | Infants Fed Mother's Own Milk | Donor Milk Fed Infants
Started | 74 | 43
Completed | 74 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infants Fed Mother's Own Milk | Donor Milk Fed Infants | Total
Number analyzed (Participants) | 74 | 43 | 117
Age, Customized [Mean (Standard Deviation); unit: weeks]
  Gestational age | 28.7 (2.0) | 28.4 (2.5) | 28.6 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 18 | 53
  Male | 39 | 25 | 64

OUTCOME MEASURES:

1. Primary Outcome: Intestinal Microbiome Diversity
Description: Stool samples during the first 6 weeks of life will be analyzed to compare development of microbial diversity
Time Frame: 6 weeks
Population: Stool samples were selected for microbiota analysis from infants who had samples collected at every time point over the first 6 weeks of life (n=90).
Measure: Mean (Standard Error); unit: taxa represented
Arm/Group | Infants Fed Mother's Own Milk | Donor Milk Fed Infants
Number analyzed (Participants) | 58 | 32
taxa represented | 55.7 (3.6) | 46.3 (4.1)

2. Primary Outcome: Hospital Length of Stay
Description: Hospital length of stay will be calculated from birth to discharge of infant.
Time Frame: Birth to discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Infants Fed Mother's Own Milk | Donor Milk Fed Infants
Number analyzed (Participants) | 74 | 43
days | 72.5 (33.2) | 88.2 (62.2)

3. Primary Outcome: Weight Gain
Description: Weight gain will be evaluated weekly throughout the study (defined as g/kg/day)
Time Frame: 6-10 weeks
Measure: Mean (Standard Deviation); unit: g/kg/day
Arm/Group | Infants Fed Mother's Own Milk | Donor Milk Fed Infants
Number analyzed (Participants) | 74 | 43
g/kg/day | 13.6 (2.2) | 12.5 (1.5)

4. Primary Outcome: Linear Growth
Description: Linear growth will be measured weekly (defined as cm/week)
Time Frame: 6-10 weeks
Measure: Mean (Standard Deviation); unit: cm/week
Arm/Group | Infants Fed Mother's Own Milk | Donor Milk Fed Infants
Number analyzed (Participants) | 74 | 43
cm/week | 1 (0.23) | 1 (0.22)

5. Primary Outcome: Head Circumference Growth
Description: Growth in head circumference will be measured weekly (defined as cm/wk)
Time Frame: 6-10 weeks
Measure: Mean (Standard Deviation); unit: cm/week
Arm/Group | Infants Fed Mother's Own Milk | Donor Milk Fed Infants
Number analyzed (Participants) | 74 | 43
cm/week | 0.8 (0.19) | 0.8 (0.17)

6. Secondary Outcome: Days to Final Enteral Feed Volume
Description: Number of days for infant to reach full enteral feeds.
Time Frame: 6-10 weeks
Population: Infants in both groups
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Infants Fed Mother's Own Milk | Donor Milk Fed Infants
Number analyzed (Participants) | 74 | 43
days | 12.4 (4.5) | 13.9 (7.0)

7. Secondary Outcome: Rates of Necrotizing Enterocolitis (NEC)
Description: the number of patients with a diagnosis of NEC (Stage ≥ IIA) will be collected
Time Frame: 6-10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Infants Fed Mother's Own Milk | Donor Milk Fed Infants
Number analyzed (Participants) | 74 | 43
Participants | 1 | 2

8. Secondary Outcome: Rates of Spontaneous Intestinal Perforation (SIP)
Description: the number of patients who develop a spontaneous intestinal perforation will be collected
Time Frame: 6-10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Infants Fed Mother's Own Milk | Donor Milk Fed Infants
Number analyzed (Participants) | 74 | 43
Participants | 0 | 2

9. Secondary Outcome: Rates of Late-onset Sepsis
Description: the number of patients with late-onset sepsis will be collected
Time Frame: 6-10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Infants Fed Mother's Own Milk | Donor Milk Fed Infants
Number analyzed (Participants) | 74 | 43
Participants | 4 | 6

ADVERSE EVENTS:
Time Frame: Through study completion (1 year).
Arm/Group | Infants Fed Mother's Own Milk | Donor Milk Fed Infants
All-Cause Mortality (participants affected / at risk) | 2/74 | 2/43
Serious Adverse Events (participants affected / at risk) | 14/74 | 20/43
Other Adverse Events (participants affected / at risk) | 26/74 | 17/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infants Fed Mother's Own Milk (N=74) | Donor Milk Fed Infants (N=43)
Necrotizing Enterocolitis (NEC)- Stage ≥ IIA (Gastrointestinal disorders) | 1 | 2 — Overall necrotizing enterocolitis (NEC) Stage ≥ IIA among study infants (all exclusively human milk-fed): 2.4% (1.6% surgical NEC).
Spontaneous Intestinal Perforation (SIP) (Gastrointestinal disorders) | 0 | 2
Late-onset sepsis (Infections and infestations) | 4 | 6
Severe bronchopulmonary dysplasia (BPD) (Respiratory, thoracic and mediastinal disorders) | 8 | 11 — Positive pressure or FiO2 > 30% at 36 wk PMA
death (General disorders) | 2 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infants Fed Mother's Own Milk (N=74) | Donor Milk Fed Infants (N=43)
BPD (Respiratory, thoracic and mediastinal disorders) | 26 | 17 — FiO2 > 21% for ≥28 d

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes